CLINICAL TRIAL: NCT06633341
Title: A Clinical Study on the Safety and Effectiveness of Targeting CD5 CAR-T Cells in the Treatment of r/r CD5+ T-lymphoma
Brief Title: Targeting CD5 CAR-T Cells in the Treatment of r/r CD5+ T-lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024013
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: T-lymphoblastic Lymphoma
Keywords: CD5 CAR-T
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD5+ T-lymphoma Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD5 CAR T-cells

INTERVENTIONS:
Biological: CD5 CAR T-cells — Each subject receive CD5+ T-lymphoma Targeted CAR T-cells by intravenous infusion
  Other Names: CD5+ T-lymphoma Targeted CAR T-cells injection

SUMMARY:
A Clinical Study on the Safety and Effectiveness of targeting CD5 CAR-T Cells in the treatment of r/r CD5+ T-lymphoma

DETAILED DESCRIPTION:
In this study, 30 patients with relapsed refractory T-lymphoma were proposed to undergo CD5 CAR-T Cells therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of CD5 CAR-T Cells therapy for relapsed refractory T-lymphoma; At the same time, on the basis of expanding the sample size, more safety data on CD5 CAR-T Cells treatment for relapsed refractory T-lymphoma were accumulated.

ELIGIBILITY:
Inclusion Criteria:

* 1. According to the 2016 WHO classification of lymphocyte tumors, histologically confirmed CD5-positive T-cell non-Hodgkin lymphoma (T-NHL),

R/R T-NHL(meets one of the following conditions) :

1. Subjects did not go into remission or relapse after receiving second-line or more chemotherapy regiments;
2. Primary drug resistance;
3. Relapse after autologous hematopoietic stem cell transplantation;

   * 2.CD5 expression rate was >90%;
   * 3. According to Lugano 2014, there should be at least one evaluable tumor lesion;
   * 4. Total bilirubin ≤51 (mol/L), Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) ≤ 3 times the upper limit of the normal range, creatinine ≤176.8 (mol/L);
   * 5. Echocardiography showed left ventricular ejection fraction (LVEF) ≥50%;
   * 6. Refers to the pulse oxygen saturation 92% or higher oxygen (state);
   * 7. Estimated life expectancy of minimum of 12 weeks;
   * 8. ECOG 0-2;
   * 9. Pregnant/lactating women, or male or female patients who have fertility and are willing to take effective contraceptive measures at least 6 months after the last cell infusion during the study period;
   * 10. Those who voluntarily participated in this trial and provided informed consent;

Exclusion Criteria:

* 1. History of epilepsy or other central nervous system disorders;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* 3. Active infection of hepatitis B virus, C virus or hepatitis E virus;
* 4. Active infected persons who are not cured;
* 5. Before using any gene therapy products;
* 6. Received anti-tumor therapy before infusion, should meet the following any one should be ruled out:

  1. treated with systemic corticosteroids therapy within 72 hours (except glucocorticoid physiological replacement therapy, such as prednisone < 10 mg/d or an equivalent dose of the drug);
  2. received within 72 hours of small molecule targeted therapy;
  3. 2 weeks received systemic chemotherapy except (pretreatment);
  4. four weeks received radiotherapy;
* 7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8. Any unsuitable to participate in this trial judged by the investigator;
* 9. Any situation that researchers believe may increase the risk to the subjects or interfere with the trial results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate ,ORR | Up to 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Progression Free Survival, PFS | Up to 2 years after Treatment
  The time from randomization or start of study treatment until objective tumor progression or death
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China